CLINICAL TRIAL: NCT03260738
Title: Preliminary Feasibility Study of Rehabilitation by Robot "Coach" of Chronic Low Back Pain Patient
Brief Title: Robot Coach of Chronic Low Back Pain Patient
Acronym: RCOOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 29BRC17.0084
Record Dates: First submitted 2017-08-08; First posted 2017-08-24 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Rehabilitation; Robot Poppy
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Robot Poppy" group (Experimental): 30 minutes of daily rehabilitation program (physical exercises dedicated to the mobility of the spine) supervised by Poppy robot during 3 weeks included in a 3hours daily (5 days a week) rehabilitation program.
  Interventions: Device: Rehabilitation program with Poppy robot
- Control group (Active Comparator): Usual 3hours daily (5 days a week) rehabilitation program without robot during 3 weeks
  Interventions: Other: Usual rehabilitation program

INTERVENTIONS:
Device: Rehabilitation program with Poppy robot — Patient with a chronic low back pain. Usual 3 hours rehabilitation daily program, 5 days a week, 3 weeks. Among those 3 hours, patients receive 30 minutes of physical exercises dedicated to mobility of the spine supervised by robot Poppy.
  Arms: "Robot Poppy" group
Other: Usual rehabilitation program — Patient with a chronic low back pain. Usual 3 hours rehabilitation daily program, 5 days a week, 3 weeks.
  Arms: Control group

SUMMARY:
The objective of KERAAL technological project is to create a new intelligent robot which allows a humanoid robot to record then to show and to follow the progress of rehabilitation sessions proposed by a physiotherapist to a patient, the latter being able to practice without the physiotherapist. The final objective is to stimulate and increase the overseen time of rehabilitation. Poppy robot was chosen as it is able to realize all kind of movements notably movements of the spine with 5 degrees of freedom associated to the several levels of the spine. It will allow to address the population included in the protocol. RCOOL study tries to validate this prototype device as tool of rehabilitation.

The main objective is the feasibility of the supervision by a humanoid robot of a succession of rehabilitation exercises.

RCOOL study is a randomized clinical trial checked under single-blind condition to compare two rehabilitation strategies, one with exercises executed by the patients and supervised by Poppy and the other one with usual rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low back pain (more than 6 months)
* Patient who has completed an outpatient rehabilitation program with at least 20 spine-centric sessions
* Inclusion in a low back pain rehabilitation program in an inpatient our outpatient unit.
* Adult between 18 and 70 years old
* Patient affiliated to French social security system
* Patient having signed an informed consent of participation for research

Exclusion Criteria:

* Symptomatic low back pain (identified medical etiology)
* Isolated sciatica, whatever the cause
* Cruralgia
* Chronic widespread pain
* Age lower than 18 and higher than 70
* Unfit of agreeing or refusing to participate in the study
* Unstable medical situation preventing the continuous realization of a program of at least 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Average time of the daily physical activity | Day 0 to Week 4
  Each therapist note the time of each physical activity session with the usually breaks. The time of kinesitherapy included the activity supervised by poppy will allow to evaluate the prototype device feasibility.

SECONDARY OUTCOMES:
Visual Analog Scale (EVA) of lumbar pain | Day 0, Week 4 and Month 6
Roland-Morris questionnaire | Day 0, Week 4 and Month 6
Dallas questionnaire | Day 0, Week 4 and Month 6
Fear Avoidance and Belief Questionnaire (FABQ) | Day 0, Week 4 and Month 6
Number of adverse events | Day 0 to Day 90
Acceptability questionnaire | Week 4 and Month 6
Number of exercises done during rehabilitation supervised by robot Poppy (30 minutes each day for 4 weeks) | Day 0 to Week 4

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - Fondation ILDYS - Service de MPR de l'appareil locomoteur de PERHARIDY, Roscoff